CLINICAL TRIAL: NCT04002193
Title: Pleth Variability Index as Predictors of Fluid Responsiveness in Modified Prone Position(Concord Position) or Knee-chest Position
Brief Title: Pleth Variability Index in Modified Prone Position or Knee-chest Position (Concord Position)
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Heesun Park, Clinical instructor of Anesthesiology and Pain department, Asan Medical Center
Other Study IDs: HePark
Record Dates: First submitted 2019-05-24; First posted 2019-06-28 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Fluid Responsiveness; Modified Prone Position
Keywords: Pleth variability index
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: volume expansion — To assess fluid responsiveness
  Other Names: If stroke volume of FloTrac® decrease 15 % of baseline, crystalloid loading of 4ml/kg will start.

SUMMARY:
To investigate whether PVI predicts the fluid responsiveness in modified prone position undergoing posterior approach cervical operation. Furthermore, modified prone position could influence on dynamic variables including stroke volume variation(SVV), pulse pressure variation(PPV) and PVI.

DETAILED DESCRIPTION:
Objective :

To compare measurements of pleth variability index (PVI), pulse pressure variation (PPV) and stroke volume variation (SVV) to predict fluid responsiveness in modified prone position or knee-chest position (concord position) for cervical operation.

To identify Influence of the modified prone position (concord position) on these variables.

Method

1. To assess influence of the position change on PVI and other variables(PPV, SVV)
2. To assess PVI to predict fluid responsiveness at modified prone position

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists'(ASA) physical status 1-3
* patients who received cervical operation in modified prone position or knee-chest position

Exclusion Criteria:

* Valvular heart disease
* Congestive heart failure, reduced left ventricular function ( Ejection fraction < 40%)
* Moderate grade of pulmonary disease
* Arrhythmia (atrial fibrillation, atrial flutter.. etc.)
* body mass index > 30 or < 15 kg/m2

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received cervical operation at modified prone position (concord position)
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
To assess influence of the position change on PVI and other variables(PPV, SVV) | 1.supine position : 5 minute after anesthesia induction with arterial-line insertion 2. 5 min after crystalloid 4 ml/kg loading / 3. modified prone position (baseline)
  When position change from supine to modified prone position, to assess the change of PVI and other variables. The correlation of PVI and cardiac output during this change.

SECONDARY OUTCOMES:
To measure dynamic variables (pulse pressure variation, stroke volume variation and pleth variability index) in modified prone position | 1. Supine position : 5 minute after anesthesia induction with arterial-line insertion 2. 5 minute after a position change to prone 3. before and after fluid loading
  Record the data of variables after 5 minute hemodynamic stability without changes of drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
We did not have the permission of data share from institutional review board.